CLINICAL TRIAL: NCT06320691
Title: General vs Spinal Anesthesia for Total Joint Arthroplasty-Anterior Approach: A Single-Institution Observational Study
Status: Completed | Type: Observational
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Sponsor
Other Study IDs: BezmialemVU 1
Record Dates: First submitted 2024-02-12; First posted 2024-03-20 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Arthroplasty Complications; Anesthesia
Keywords: total hip arthroplasty; general anesthesia; spinal anesthesia; direct anterior approach
MeSH Terms: interventions — Arthroplasty, Replacement, Hip; Anesthesia, General; Anesthesia, Spinal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- General Anesthesia Group: The group that underwent direct anterior total hip arthroplasty with general-systemic anesthesia
  Interventions: Procedure: Total Hip Arthroplasty; Procedure: General Anesthesia
- Spinal Anesthesia Group: The group that underwent direct anterior total hip arthroplasty with spinal-neuraxial anesthesia
  Interventions: Procedure: Total Hip Arthroplasty; Procedure: Spinal Anesthesia

INTERVENTIONS:
Procedure: Total Hip Arthroplasty — Patients that underwent direct anterior approach total hip arthroplasty
Procedure: General Anesthesia — Patients that underwent general/systemic anesthesia before surgery
  Groups: General Anesthesia Group
Procedure: Spinal Anesthesia — Patients that underwent spinal/neuraxial anesthesia before surgery
  Groups: Spinal Anesthesia Group

SUMMARY:
The study compares the effects of various anesthetic techniques on anterior approach total hip arthroplasty results retrospectively

DETAILED DESCRIPTION:
Under general (GA) or spinal anesthesia (SA), total hip arthroplasty using the anterior approach (THA-A) can be safely performed. The best method is not sufficiently described in the literature currently in existence.This observational study was carried out at a single facility with consecutive enrollment of patients getting primary THA-A. The investigators compared the difference in complication rates, intraoperative blood loss, length of hospital stay, and duration of surgery, acetabular and femoral component orientation and stem subsidence.

ELIGIBILITY:
Inclusion Criteria:

* patients who underwent direct anterior approach primary total hip arthroplasty with general anesthesia
* patients who underwent direct anterior approach primary total hip arthroplasty with spinal anesthesia

Exclusion Criteria:

* patients who underwent revision total hip arthroplasty
* patients who underwent total hip arthroplasty with approaches other than direct anterior approach
* patients who underwent primary total hip arthroplasty due to hip fractures

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: - patients who underwent direct anterior approach primary total hip arhtroplasty with hip osteoarthritis
Sampling Method: Probability Sample
Enrollment: 437 (Actual)
Dates: Start 2014-01-10 (Actual); Primary Completion 2017-01-10 (Actual); Study Completion 2017-05-25 (Actual)

PRIMARY OUTCOMES:
Mean intraoperative estimated blood loss | from preoperative session to postoperative 1 day
  Total blood volume was calculates according to Nadler's formula based on patient's sex, height and weight of the patient, whereas the estimated blood loss was calculated according to Meunier's formula (mL)
mean duration of surgery | from preoperative session to postoperative 1 day
  Duration of total hip arthroplasty surgery for each patient
length of hospital stay | from the date of total hip arthroplasty operation until the day that patients discharge, assesed up to 7 days
  from date of operation until the date of discharge
stem subsidence | postoperative 1 year
  Subsidence was evaluated by comparing immediate post-operative radiographic images with those obtained at 1 year follow-up. Subsidence was measured as a vertical drop of stem, characterised by a radiolucent line at the proximal most aspect of the bone-prosthesis interface.
stem varus/valgus degrees | postoperative 1 year
  varus or valgus angulation of femoral stem after surgery
acetabular abduction | postoperative 1 year
  abduction degree of acetabular component after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Bezmialem Vakif University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided